CLINICAL TRIAL: NCT01646723
Title: Volunteers Adding Life in Dementia (VALID)
Brief Title: Volunteers Adding Life in Dementia
Acronym: VALID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Dallas Seitz, MD, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VALID1
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Alzheimer Disease; Behavior
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavior | interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VALID Intervention (Experimental): Volunteers Adding Life in Dementia (VALID) Program
  Interventions: Behavioral: Volunteers Adding Life in Dementia (VALID) Program

INTERVENTIONS:
Behavioral: Volunteers Adding Life in Dementia (VALID) Program — The VALID intervention will consist of 2 phases. First, volunteers will complete an assessment involving recording of a "Life Story" for each patient participant. This will include information on the patient's psychosocial history, occupational history, hobbies, interests and preferred activities using information from the LTC medical record and interviews with the patient and family members. Based on this information, a variety of potential psychosocial interventions will be developed for the individual with the assistance of the recreation therapist at the LTC. The second phase will involve implementation of the VALID intervention. Each individual with dementia will receive personalized pleasant activities for a minimum session of 30 minutes at a frequency of 3 times per week. One volunteer will complete the "Life Story" assessment and up to 3 volunteers may be involved with implementing the VALID program for each resident.

SUMMARY:
The objectives of our project are to: 1.) Develop a training program and manual for volunteers to implement evidence-based, non-pharmacological interventions for neuropsychiatric symptoms (NPS) of dementia in long-term care (LTC) settings; 2.) Recruit and train volunteers using the VALID program and pilot test the volunteer-led program with 20 individuals with Alzheimer's disease and NPS in a LTC facility in Kingston; and, 3.) Evaluate the effects of the VALID program on the symptoms of NPS, patient quality of life, volunteer's experience, and LTC staff stress.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Alzheimer's disease or related forms of dementia
* significant symptoms of agitation as measured by a Cohen-Mansfield Agitation Inventory (CMAI) total score of >39
* in nursing home for at least 30 days
* presence of a caregiver or substitute decision maker willing to consent to treatment
* no changes in psychotropic medications in the 2 weeks preceding enrolment in study

Exclusion Criteria:

* depressive symptoms presenting risk
* physically aggressive behavior posing safety risk to others
* uncontrolled pain
* currently receiving palliative care
* medically unstable with life expectancy of < 6 months
* currently awaiting transfer to another LTC facility or hospital.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Cohen-Mansfield Agitation Inventory (CMAI) score | Baseline and 12 weeks

SECONDARY OUTCOMES:
Clinically significant reduction in agitation | Baseline and 12 weeks
  30% reduction in CMAI score
Remission of neuropsychiatric symptoms | Baseline and 12 weeks
  CMAI score <40
Change in Neuropsychiatric Inventory (NPI) score | Baseline and 12 weeks
Change in depression symptoms (Cornell Depression in Dementia Rating Scale) | Baseline and 12 weeks
Dementia Quality of Life (DemQoL) Scale | Baseline and 12 weeks
Clinical Global Impression of Change (CGI-C) | Baseline and 12 weeks
Use and dose of required medication | Baseline and 12 weeks
Short form health survey | Baseline and 12 weeks
  Volunteer quality of life
Change in Modified Nursing Care Assessment Scale score | Baseline and 12 weeks
  Assessing nursing stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dallas P Seitz, MD, Principal Investigator — Queen's University
Locations (1):
- Extendicare Kingston, Kingston, Ontario, Canada